CLINICAL TRIAL: NCT00003832
Title: Cell Kinetic Study of Bromodeoxyuridine (BrdU) in Prostate Cancer
Brief Title: Broxuridine Plus Surgery in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02297; 98-374; CDR0000066989 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-09-30 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bromodeoxyuridine; 5-bromouridine; Surgical Procedures, Operative; Congresses as Topic

ARMS (1):
- Treatment (bromodeoxyuridine) (Experimental): Patients receive broxuridine IV over 30 minutes on day -1. Approximately 12-96 hours later, patients undergo surgery to remove the prostate.Tumor tissue is examined by immunostaining for the presence of broxuridine to determine doubling times of the tumor.
  Interventions: Drug: bromodeoxyuridine; Procedure: conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bromodeoxyuridine — Given IV
  Other Names: 5-BrdU; 5-bromodeoxyuridine; BrdU; broxuridine
Procedure: conventional surgery — Undergo surgery
  Other Names: surgery, conventional
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of broxuridine in treating patients who are undergoing surgery for stage I or stage II prostate cancer. Broxuridine may help doctors determine the rate of growth of prostate tumors and help them plan effective treatment

DETAILED DESCRIPTION:
OBJECTIVES:

I. Measure the potential doubling times of multifocal adenocarcinomas of the prostate using broxuridine.

II. Determine whether the doubling times of multifocal carcinomas occurring within a single prostate are consistent with a model in which low-volume carcinomas have slow doubling times and high-volume carcinomas have fast doubling times.

OUTLINE:

Patients receive broxuridine IV over 30 minutes on day -1. Approximately 12-96 hours later, patients undergo surgery to remove the prostate. Tumor tissue is examined by immunostaining for the presence of broxuridine to determine doubling times of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I or II (T1-2) carcinoma of the prostate

  * PSA greater than 8 ng/mL
  * Abnormal findings on digital rectal examination
* Eligible for radical prostatectomy
* Performance status - ECOG 0 or 1
* No prior biologic therapy
* No prior chemotherapy
* No prior neoadjuvant hormonal therapy
* No prior radiotherapy
* See Disease Characteristics
* No prior therapy that would affect tumor growth rates or volume

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1999-07; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Average doubling time between low and high volume tumors | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Glode, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States